CLINICAL TRIAL: NCT01547078
Title: A Phase 2 Clinical Study of Lyophilized Plasma in Patients With Acquired Coagulopathy Due to Liver Disease
Brief Title: Clinical Study of Lyophilized Plasma in Patients With Liver Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-I-LyP-2
Record Dates: First submitted 2012-02-10; First posted 2012-03-07 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Liver Disease
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Licensed Plasma (Active Comparator)
  Interventions: Biological: Licensed Plasma
- Lyophilized Plasma (Experimental)
  Interventions: Biological: Lyophilized Plasma

INTERVENTIONS:
Biological: Lyophilized Plasma — Licensed plasma that has been lyophilized.
  Arms: Lyophilized Plasma
Biological: Licensed Plasma — Plasma that has been authorized for transfusion.
  Arms: Licensed Plasma

SUMMARY:
A multi-center, phase 2, randomized, controlled study of the effect of lyophilized plasma in patients with liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years of age.
2. Patients with liver disease.
3. Patients who have need for plasma therapy for a surgical or an invasive procedure or who have evidence of bleeding.
4. Patients with an elevated international normalized ratio due to liver disease.
5. Patients who have given written informed consent or for whom written informed consent has been obtained from the patient's legal representative on their behalf.
6. Patients able and willing to comply with the procedures laid out in the study protocol.

Exclusion Criteria:

1. Patients who are clinically unstable.
2. Patients who have received mediations that could interfere with results of laboratory testing.
3. Patients who have congenital or acquired coagulopathies of non-hepatic origin.
4. Pregnant or nursing women.
5. Active illicit drug use.
6. Patients participating in another clinical treatment study currently or during the past 1 month prior to study inclusion.
7. Patients previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Assess and compare adverse events | Duration of Study (Less than or equal to 7 days)
  The primary safety objective is to assess the incidence of adverse events of lyophilized plasma compared to control.